CLINICAL TRIAL: NCT06608524
Title: Effect of Self-regulated Learning on Academic Performance Among Physical Education Students in Shanxi, China
Brief Title: Effect of Self-regulated Learning on Academic Performance Among Physical Education Students
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: XIE HUIJUAN (Other)
Responsible Party: Sponsor-Investigator, XIE HUIJUAN, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KL202403
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Academic Performance
Keywords: self-regulated learning; academic performance; physical education

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group will use self-regulated learning strategy, and the control group will use standard learning method. Each parallel group has 40 physical education stuednts.
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group used self-regulated learning strategy to improve academic performance of physical education students in China.
  Interventions: Behavioral: Self-regulated learning strategy
- Control group (Active Comparator): The control group used standard learning method to improve physical education academic performance.
  Interventions: Behavioral: Standard learming method

INTERVENTIONS:
Behavioral: Self-regulated learning strategy — The experimental group uses self-regulated strategy.This program selects classroom performance , homework quality , experimental operation, and test score as academic performance (score) evaluation variables.
  Arms: Experimental group
Behavioral: Standard learming method — The control group uses standard learming method. The program selects classroom performance, homework quality, experimental operation, and test score evaluation form as academic performance (score) evaluation variables.
  Arms: Control group

SUMMARY:
Difficulty in employment for college students is a serious social problem in China. All qualification examinations, further education and jobs require written theory tests. Many students are affected by their examinations, additional studies, and employment due to poor academic performance and insufficient learning ability. College students majoring in physical education generally perform better in motor technical skills but often encounter difficulties in theoretical learning.

According to the existing literature and many studies, self-regulated learning is an advanced form of metacognitive learning (Pintrich, 2004). It helps cultivate students' independent learning ability and can improve their theoretical academic performance. This study attempts to use self-regulated learning in physical education theory classes to examine whether this method can enhance physical education students' theoretical academic performance.

DETAILED DESCRIPTION:
In this study, the experimental group received a 12-week (John, 2017) self-regulated learning strategy based on a learning model teaching intervention designed for this study. In contrast, the control group discussed and studied traditional learning content for 12 weeks with the teacher, and the students in the experimental group learned the self-regulated learning strategy. A cluster-randomised controlled trial (CRCT) design was used, and the experimental and control groups were randomly assigned to two schools. After 12 weeks of learning, both groups were required to conduct a learning performance assessment.

ELIGIBILITY:
Inclusion Criteria:

1. University students;
2. Major in Physical Education;
3. Health;
4. Able to attend all evaluation;
5. Understand the study purposes and procedures;
6. No previous experience performing self-regulated learning strategy.

Exclusion Criteria:

1. University students not majoring in Physical Education;
2. Exclude participants who have not finished all evaluation;
3. Not understanding the study purposes and procedures;
4. Participants with an experience in self-regulated learning strategy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Class Performance Evaluation Form | Pretest: Before experiment; Post-test: 12 weeks end.
  A form is used to evaluate the physical education students' academic performance when the teacher uses class performance evaluation form.
Homework Quality Evaluation Form | Pretest: Before experiment; Post-test: 12 weeks end.
  A form is used to evaluate the physical education students' academic performance when the teacher uses homework quality evaluation form.
Experimental Operation Evaluation Form | Pretest: Before experiment; Post-test: 12 weeks end.
  A form is used to evaluate the physical education students' academic performance when the teacher uses experimental operation evaluation form.
Test Score Evaluation Form | Pretest: Before experiment; Post-test: 12 weeks end.
  A form is used to evaluate the physical education students' academic performance when the teacher uses test score evaluation form.
Academic Performance (Score) Evaluation Form | Pretest: Before experiment; Post-test: 12 weeks end.
  A form is used to evaluate the physical education students' academic performance when the teacher uses academic performance (score) evaluation form.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuncheng University, Yuncheng, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.Davis, L. L. (1992). Instrument review: Getting the most from a panel of experts. Applied nursing research, 5(4), 194-197. 2.Goudas, M., Dermitzaki, I., & Kolovelonis, A. (2017) Self-regulated learning and students' metacognitive feelings in physical education. International Journal of Sport and Exercise Psychology, 15(2), 131-145. 3. John Sproule(2017). Physical education in Taiwan: when students begin to take control. International Sport Studies, 39(1): 1-18. 4. Pintrich PR(2004). A conceptual framework for assessing motivation and self-regulated learning in college students. Educational Psychology Review 16(4): 385-407. 5. Rosenkranz, R. R., Lubans, D. R., Peralta, L. R., Bennie, A., Sanders, T., & Lonsdale, C. (2012). A cluster randomized controlled trial of strategies to increase adolescents' physical activity and motivation during physical education lessons: The motivating active learning in physical education (MALP) trial. BMC Public Health, 12, 834. doi:10.1186/1471-2458-12-834 6. Zamanzadeh, V., Ghahramanian, A., Rassouli, M., Abbaszadeh, A., Alavi-Majd, H., & Nikanfar, A. R. (2015). Design and implementation content validity study: development of an instrument for measuring patient-centered communication. Journal of caring sciences, 4(2), 165. 7. Zimmerman, B. J. (1990). Self-regulated learning and academic achievement: An overview. Educational Psychologist, 25(1), 3-17. 8. Zimmerman, B. J. 2000. "Attaining Self-Regulation: A Social-Cognitive Perspective." In Boekaerts, M., Pintrich P., and Zeidner M. (Eds.), Self-regulation: Theory, Research, and Applications, Academic, Orlando, FL: 13-39. 9. Zimmerman, B. J. (2001). Theories of self-regulated learning and academic achievement: An overview and analysis. In B. J. Zimmerman, & D. H. Schunk (Eds.), Self-regulated learning and academic achievement: Theoretical perspectives (pp. 1-37). Mahwah, NJ: Erlbaum.